CLINICAL TRIAL: NCT02361489
Title: Clinical Study to Compare Various Dosing and Titration Guidelines of Insulin Delivered Via V-Go ® in Patients With Type 2 Diabetes Initiating Basal Bolus Therapy in Primary Care Offices (Short Title: TITRATE)
Brief Title: Clinical Study to Compare Various Dosing and Titration Guidelines of Insulin Delivered Via V-Go ® in Patients With Type 2 Diabetes Initiating Basal Bolus Therapy in Primary Care Offices
Acronym: TITRATE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Valeritas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSP-029
Record Dates: First submitted 2015-02-06; First posted 2015-02-11 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Titration Algorithm A (Active Comparator): All patients that are initiated on a V-Go 20 will have a starting bolus dose of 6 clicks (12 units) during the day and all patients who are initiated on a V-Go 30 will have a starting bolus dose of 9 clicks (18 units) during the day. All patients randomized to Algorithm A will use a fixed starting dose of either 2 clicks per meal (if on the V-Go 20) or 3 clicks per meal (if on the V-Go 30).
  Interventions: Device: V-Go
- Titration Algorithm B (Active Comparator): All patients that are initiated on a V-Go 20 will have a starting bolus dose of 6 clicks (12 units) during the day and all patients who are initiated on a V-Go 30 will have a starting bolus dose of 9 clicks (18 units) during the day. All patients randomized to Algorithm B will have 50% of their initial bolus dose given at the largest meal with less bolus insulin at the other meals as noted below:
  Interventions: Device: V-Go

INTERVENTIONS:
Device: V-Go — Initiation and titration of V-Go® using one of two dose titration algorithms to achieve improved A1C at 4 months.

SUMMARY:
The aim of the study is to observe patients with Type 2 Diabetes on basal insulin alone or basal insulin with oral agents can be efficiently and safely started with meal time insulin using U100 rapid acting insulin analog and V-Go® Disposable Insulin Delivery Device (V-Go) using one of two dose titration algorithms to achieve improved A1C at 4 months.

DETAILED DESCRIPTION:
This study addresses the informational needs of Primary Care Physicians with regard to providing insulin dosing and titration information utilizing a V-Go disposable insulin delivery device. We look to compare two treatment arms of insulin dosing and titration in patients with Type 2 insulin-dependent diabetes - a fixed dose titration arm, and an arm where 50% of the insulin dose is given at the largest meal of the day. This study will provide practical information on glycemic control, dose requirements and safety in patients with Type 2 diabetes on basal insulin with or without oral anti-diabetic agents who are being primarily managed in the primary care office.

ELIGIBILITY:
Inclusion Criteria: Patients must meet all of the following inclusion criteria to be eligible for enrollment into the study:

* Age ≥ 21 and ≤80 at time of study enrollment
* Ability to read and understand English
* BMI ≥ 25 kg/m2
* Weight less than or equal to 300 pounds.
* A1C ≥8 but ≤12% (most recent value within 4 weeks of baseline visit)
* Currently using any basal insulin therapy (NPH, Levemir, Lantus) with total daily dose of 30 to 120 units, and where basal dose is greater than the patient's BMI #
* Willing to attend their physician's office for follow-up visits
* Willing and able to understand and sign a written informed consent form (ICF) indicating that they agree to participate and have been informed of all pertinent aspects of the study
* Must be willing to take and record at least 3 glucose measurements per time period (pre-breakfast, lunch, dinner and bed) per week.
* Willing to opt-in into Valeritas Customer Care so that they can receive device support and reminders throughout the study
* Most recent primary care office visit at one of the participating sites.

Exclusion Criteria:Patients presenting with any the following exclusion criteria will not be eligible for enrollment into the study:

* Patient with confirmed Type 1 diabetes and/or patients with a weight greater than 300 lbs.
* Diagnosis of an Autoimmune disease affecting metabolism
* Currently using GLP-1 medications
* Current (within the last 6 months) or planned use of insulin pump for diabetes management or the use of U500 insulin.
* Ongoing participation in any clinical study
* Pregnant, lactating or intending to become pregnant
* Current chronic systemic steroid use
* Prior V-Go use

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
A1C | 4 months
  Change change in A1C from baseline (randomization) to endpoint (approximately 16 weeks).

SECONDARY OUTCOMES:
Change in glycemic control | 4 months
  • Difference in the change from baseline (randomization) to end of study visit at 4 months on glycemic control (as measured by A1C level) between the two treatment groups in a pragmatic clinical practice setting
Patient Treatment Satisfaction | 4 months
  • Between-group and within-group differences (baseline to end of study visit at 4 months) in patient treatment satisfaction in adult Type 2 patient with diabetes in a real world setting
Insulin Dose | 4 months
  • Total daily dose of insulin from baseline to end of study and to evaluate the between-group and within-group differences between the two dosing and titration arms
A1c at goal | 4 months
  Percentage of patient achieving a A1C of ≤7%
7 point glucose profile | 4 months
  Capture and analyze seven-point glucose profile at baseline and end of study
Hypoglycemia | 4 months
  Rates of hypoglycemic events and utilization

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Harris, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Wilkes-Barre, Pennsylvania, United States